CLINICAL TRIAL: NCT00606957
Title: The Effect of Vitamin D Repletion on Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Allegra Grossman, MD, The Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUH IRB# AGR-0623
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: Obesity; Metabolism
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — Vitamin D will be taken orally, 10,000 IU (0.25 mg) three times per week.

SUMMARY:
The reason for doing this study is to learn whether raising a person's vitamin D level from below normal to normal levels will improve his or her body's ability to use sugar. Vitamin D is well known to be an important vitamin for the development and maintenance of bones. Recently, scientists have learned that vitamin D may have a role in the prevention of cancer, diabetes, and autoimmune diseases. The investigators are specifically interested in studying this question in the overweight/obese population as they are at greater risk for both vitamin D deficiency and impaired ability to metabolize sugar (glucose intolerance).

Primary Hypotheses:

Vitamin D repletion (increasing the serum 25(OH)D level from ≤ 20 ng/ml to ≥ 30 ng/ml) will improve insulin sensitivity in individuals who are overweight/obese and insulin resistant.

Secondary Hypotheses:

1.Vitamin D repletion will improve biomarkers of cardiovascular risk and inflammation (directly altering macrophage cytokine production and/or indirectly as a result of improvement in insulin sensitivity.) 2.30,000 IU (0.25 mg) weekly of cholecalciferol (vitamin D3) will raise serum 25(OH)D levels from ≤ 20 ng/ml to ≥ 30 ng/ml overweight/obese population.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking men and women, ages 18-65
* Body mass index (BMI) ≥ 28 kg/m² and within 10% of maximum weight
* Serum 25(OH)D level ≤ 20 ng/ml
* Serum insulin level ≥ 7.2 mU/l
* Willingness to maintain current body weight for the duration of the study
* Willingness to maintain baseline lifestyle activities and routines for the duration of the study
* Willingness to avoid the use of non-steroidal anti-inflammatory drugs (NSAIDS), including low-dose daily aspirin, for at least ten days prior to each admission (due to the potential effects of these agents on inflammatory markers.)
* Willingness to avoid the use of all over-the-counter or prescription vitamins, dietary supplements, and herbal products during the study, with the exception of a basic multivitamin supplement.
* If of childbearing potential, willingness to use highly effective contraception for the duration of the study.

Exclusion Criteria:

* Current tobacco smoking
* History of bleeding or coagulation disorders
* Gastrointestinal disease resulting in significant gastrointestinal dysfunction or malabsorption
* History of diabetes, or diagnosed during screening OGTT
* Current treatment with hypertensive medications
* History of cardiovascular disease
* Renal disease, as evidenced by a serum creatinine above the upper limit of normal on more than one screening visit
* History of kidney stones
* History of chronic hepatitis, or liver enzymes (AST or ALT) more than 2.5 times the upper limit of normal
* Primary hyperparathyroidism or baseline hypercalcemia from any cause
* Current treatment with over-the-counter or prescription weight loss medications, such as orlistat or sibutramine
* History of bariatric surgery
* Current treatment with any cholesterol-lowering medications, such as statins, niacin, fibrates, or ezetimibe
* Blood pressure ≥ 145/90 after ten minutes of rest on more than one screen visit
* Hyperthyroidism or untreated hypothyroidism. Subjects with chronic, treated, stable hypothyroidism may be included in the study at the discretion of the Principal Investigator.
* Pregnancy, desired pregnancy, or lactation within the study period.
* HIV, Hepatitis B and C
* Medical conditions requiring daily calcium supplementation or antacid use
* Use of medications known to interact with calcium or vitamin D metabolism (bisphosphonates, corticosteroids, thiazide diuretics, cholestyramine, colestipol, mineral oil, phenytoin, barbituates, dititalis glycosides, antacids)
* Subjects with known hypersensitivity to cholecalciferol
* Participation in an investigational drug study within one month of screening
* History, physical, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the principal investigator, make the candidate ineligible for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is change in insulin sensitivity over time, as measured by the glucose clamp, HOMA and OGTT. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allegra Grossman, MD, Principal Investigator — The Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States